CLINICAL TRIAL: NCT03691272
Title: Treatment of Persistent Headache Attributed to Mild Traumatic Injury to the Head (PHATIH) in Patients With Persistent Post Concussion Symptoms (PPCS) Using Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: rTMS Treatment of Persistent Headache and Post Concussion Symptoms Attributed to Mild Traumatic Injury to the Head
Acronym: TOPiCS-rTMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-2377
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2018-09

CONDITIONS: Brain Injuries, Traumatic; Concussion, Brain; Headaches Chronic; Headache; Post-Traumatic Headache; Mild Traumatic Brain Injury; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Headache Disorders; Headache; Post-Traumatic Headache | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized with a random number generator to receive either sham or rTMS. Allocation will be concealed through the use of sequentially numbered, sealed, opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS- Real Air Film Coil (Experimental): Patient MR brain scans will be loaded and processed using the Brainsight TMS neuronavigation software and stereotaxic data for localization of the TMS stimulation site will be determined through a co-registration method between the TMS coil position and the projected site on the MR brain scan. The DLPFC will be located through MNI coordinates (-48, 20, 34). Electromyography (EMG) electrodes will be attached to the right abductor digiti minimi (ADM) muscle. The resting motor threshold (RMT) is determined as the minimal stimulation intensity required to elicit motor-evoked response of 50 microvolts peak-to-peak amplitude in at least 5 out of 10 consecutive trials of the ADM (contralateral to stimulation).
  Interventions: Device: rTMS - Real Air Film Coil
- rTMS- Sham coil (Sham Comparator): The same procedure for determining RMT as described above will be employed for the Sham Arm. However, a sham coil will be used when the treatment over the left DLPFC is applied.
  Interventions: Device: rTMS - Sham Coil

INTERVENTIONS:
Device: rTMS - Real Air Film Coil — 70% resting motor threshold amplitude; Frequency 10 Hz; 10 trains of 60 pulses/train (total of 600 pulses); Inter-train interval 45s.
  Other Names: Repetitive Transcranial Magnetic Stimulation
  Arms: rTMS- Real Air Film Coil
Device: rTMS - Sham Coil — A sham coil will be applied to the scalp after the resting motor threshold is determined. Patients will be able to hear the sound and feel the vibration of sham coil, but will not experience any effective stimulation.
  Arms: rTMS- Sham coil

SUMMARY:
The objective of this study is to investigate the treatment effect of repetitive transcranial magnetic stimulation in patients with a history of both persistent post-traumatic headache and post-concussion symptoms. In this double-blind, sham-controlled, concealed allocation, randomized clinical trial, 20 patients aged 18-65 yrs will be recruited from the Calgary Brain Injury Program (CBIP) and the Calgary Headache Assessment and Management Program (CHAMP) / Calgary Chronic Pain Centre, Calgary, Alberta, Canada. Patients will engage in a two-week rTMS treatment protocol (10 treatments) and will be followed for 6 months after therapy.

DETAILED DESCRIPTION:
Demographic information will be collected two weeks prior to starting the study including age, sex, education, headache history, concussion history, past medical history, medication use, and family medical history. Headache history will be collected including frequency, severity, medication-use, type of headache, associated symptoms (i.e. neck pain, photophobia, phonophobia, nausea, vomiting) and headache triggers. Baseline questionnaires will be completed including headache intensity scale - 6 (HIT-6), Rivermead PPCS questionnaire, British Columbia post-concussion symptom inventory (BC-PSI), Montreal cognitive assessment (MoCA), quality of life after brain injury questionnaire (QOLIBRI), patient health questionnaire-9 (PHQ-9), generalized anxiety disorder scale-7 (GADS-7) and the post traumatic stress disorder checklist for DSM-5 (PCL-5). Patients will keep a two-week baseline headache diary before treatment, 2 weeks during treatment, 2 weeks following rTMS, and for 2 weeks at the 1, 3, and 6 month follow up assessments (total of 12 weeks). Patients will be reassessed at the completion of their rTMS treatment (day 14), and at 1, 3, and 6 months post-treatment. The questionnaires including: HIT-6, Rivermead PPCS questionnaire, PC-PSI, QOLIBRI, PHQ-9 and GAD-7 will be completed at all follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a persistent headache attributed to traumatic injury to the head based on the ICHD-3 criteria
* Diagnosis of persistent post-concussion symptoms based on the ICD-10 criteria
* mTBI occurrence from 3 months to 5 years from study start date

Exclusion Criteria:

* Prior history of TMS therapy
* TMS-related contraindications (pacemaker, metallic implant)
* History of chronic headache (>15 days/month for 3 months) or migraine prior to most recent trauma
* Other medical conditions such as: structural brain disease, previous seizure, psychotic disorders (schizophrenia, bipolar disorder), liver or kidney disease, malignancy, uncontrolled hypertension or diabetes, and pregnancy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change in headache severity from baseline to 1 month post-treatment. | Repeated measures: Baseline (0-2 weeks),1 month (6-8 weeks)
  Numeric Pain Rating Scale (NPRS): a tool to assess severity of pain, which is graded from 0-10 (11 points) with 0 defined as "no pain" and 10 as "worst possible pain".
Change in headache frequency from baseline to 1 month post-treatment. | Repeated measures: Baseline (0-2 weeks),1 month (6-8 weeks)
  Number of headaches/2 weeks

SECONDARY OUTCOMES:
Headache severity | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  Numeric Pain Rating Scale (NPRS): a tool to assess severity of pain, which is graded from 0-10 (11 points) with 0 defined as "no pain" and 10 as "worst possible pain".
Headache frequency | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  Number of headaches/2 weeks
Function | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  Headache Impact Test (HIT-6): a global measure of headache impact. Addresses the 6 categories of headache impact including social, role, and cognitive functioning, vitality, psychological distress, and severity of headache pain. Each question is scored on a 5 point scale: never, rarely, sometimes, very often, and always. Total score can range from 36-78, with higher total score indicating greater impact.
Depression | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  Patient Health Questionnaire - 9 (PHQ-9): a 9 item tool used to assess the presence and severity of depressive symptoms. Each item is rated based on the frequency of occurrence in the past two weeks and is graded on a 0-3 scale (0=not at all, 1= several days, 3= nearly every day). Finally, one question rates how difficult problems have made completing tasks at home, doing work, and getting along with people. This is graded on a 4 point scale from not difficult at all to extremely difficult. Total score is calculated out of 27, with a values indicating severity of depression (i.e. 0-4= none to mild, 5-9 = mild, 10-14 = moderate, 15-19 = moderately severe, and 20-27 = very severe).
Anxiety | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  Generalized Anxiety Disorder (GAD-7): a 7-item tool where similar to the PHQ-9, each item is rated on frequency over a 2 week period based on a 0-3 scale (0=not at all, 1= several days, 3= nearly every day). Total score GAD-7 total score ranges from 0 to 21, with scores indicating severity of anxiety (i.e. 0-5= mild, 6-10 = moderate, 11-15 = moderately severe, 16-21 = very severe).
Post-traumatic Stress Disorder | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  PTSD Checklist for DSM-5 (PCL-5): is a paper and pencil self-report measure, which rates the severity of PTSD symptoms over the past month. It is composed of 4 subscales, and is a total of 20 items long. Each item corresponds to the 20 criteria for PTSD defined in the DSM-5.
Cognition | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  Montreal Cognitive Assessment (MoCA):a paper and pencil global cognitive assessment tool which measures 7 neurocognitive domains including visuospatial/executive function, naming, memory, attention, language, abstraction and orientation. It is composed of 16 items and scored out of 30 points.
Quality of Life (QoL): QOLIBRI | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  The QOLIBRI is a health-related quality of life instrument developed specifically for patients who have experienced a traumatic brain injury. It has 6 subscales and a total of 37 items. The tool is divided into two sections. The first addresses satisfaction with health related quality of life, characterized by cognition, self, autonomy in daily life, and social aspects. These are reported on a 1-5 scale with 1 defined as "not at all satisfied" and 5 as "very satisfied". The second section is related to "feeing bothered by" emotions and physical problems. They are again scored from 1-5, however 1 is defined as "very bothered" and 5 as "not bothered at all". The score from all subscales are totaled, and then divided by the number of responses. This gives a mean score, which can range from 1-5. Next, 1 is subtracted from the mean and then multiplied by 25 to produce a score on the 0-100 scale (0=worst possible quality of life, 100= best possible quality of life).
Post-concussion Symptoms | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  Rivermead Post-concussion Symptoms Questionnaire (RPQ): an instrument developed to assess the frequency and severity of 16 common post-concussion symptoms. On this paper and pencil tool, patients rate the extent to which their symptoms (compared to their pre-injury levels) have become more problematic over the past 24 hours using a rating scale from 0-4 (0=not experienced, 1=no more of a problem, 2=mild problem, 3=moderate problem, 4=severe problem). A total symptom score is calculated out of 64.
Post-concussion Symptoms | Repeated measures: Pre-treatment (0-2 weeks), During Treatment (2-4 weeks), Post-treatment (4-6 weeks), 1 Month (6-8 weeks), 3 Months (10-12 weeks), 6 Months (22-24 weeks)
  British Columbia Post-concussion symptom inventory (BC-PSI): a 16 item instrument, where 13 questions are used to assess the frequency and intensity of post-concussion symptoms as defined by ICD-10 criteria over the past two weeks (i.e. headaches, dizziness or light-headedness, nausea, fatigue, phonophobia, sadness, nervousness or tension, temper problems, poor concentration, memory problems, reading difficulty, and sleep disturbance). Severity is rated from 0-5 (6 point scale) where 0 is defined as "not at all" and 5 as "constantly". Intensity is also rated from 0-5, where 0 is defined as "not at all" and 5 as "very severe problem". The two items are then multiplied (frequency x intensity) for each item. This is subsequently converted to item total scores where: 0-1=0, 2-3=1, 4-6=2, 8-12=3, and ≥15=4. Scores from 1-2 signify mild symptoms and ≥3 moderate to severe symptoms, which can be considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Chantel Debert, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (1):
- University Of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Misra UK, Kalita J, Bhoi SK. High-rate repetitive transcranial magnetic stimulation in migraine prophylaxis: a randomized, placebo-controlled study. J Neurol. 2013 Nov;260(11):2793-801. doi: 10.1007/s00415-013-7072-2. Epub 2013 Aug 21. PMID 23963471
- [Background] Iverson GL, Brooks BL, Ashton VL, Lange RT. Interview versus questionnaire symptom reporting in people with the postconcussion syndrome. J Head Trauma Rehabil. 2010 Jan-Feb;25(1):23-30. doi: 10.1097/HTR.0b013e3181b4b6ab. PMID 19680134
- [Background] Iverson GL, Lange RT. Examination of "postconcussion-like" symptoms in a healthy sample. Appl Neuropsychol. 2003;10(3):137-44. doi: 10.1207/S15324826AN1003_02. PMID 12890639
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Eyres S, Carey A, Gilworth G, Neumann V, Tennant A. Construct validity and reliability of the Rivermead Post-Concussion Symptoms Questionnaire. Clin Rehabil. 2005 Dec;19(8):878-87. doi: 10.1191/0269215505cr905oa. PMID 16323387
- [Background] Lannsjo M, Borg J, Bjorklund G, Af Geijerstam JL, Lundgren-Nilsson A. Internal construct validity of the Rivermead Post-Concussion Symptoms Questionnaire. J Rehabil Med. 2011 Nov;43(11):997-1002. doi: 10.2340/16501977-0875. PMID 22031345
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Ashbaugh AR, Houle-Johnson S, Herbert C, El-Hage W, Brunet A. Psychometric Validation of the English and French Versions of the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). PLoS One. 2016 Oct 10;11(10):e0161645. doi: 10.1371/journal.pone.0161645. eCollection 2016. PMID 27723815
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Lowe B, Schenkel I, Carney-Doebbeling C, Gobel C. Responsiveness of the PHQ-9 to Psychopharmacological Depression Treatment. Psychosomatics. 2006 Jan-Feb;47(1):62-7. doi: 10.1176/appi.psy.47.1.62. PMID 16384809
- [Background] Fann JR, Bombardier CH, Dikmen S, Esselman P, Warms CA, Pelzer E, Rau H, Temkin N. Validity of the Patient Health Questionnaire-9 in assessing depression following traumatic brain injury. J Head Trauma Rehabil. 2005 Nov-Dec;20(6):501-11. doi: 10.1097/00001199-200511000-00003. PMID 16304487
- [Background] Kumar, S., Jawahar, A., Shah, P. & Kumar, M. Montreal Cognitive Assessment, a screening tool for Mild Traumatic Brain Injury (P7.185). Neurology 84 (2015).
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Kjeldgaard D, Forchhammer H, Teasdale T, Jensen RH. Chronic post-traumatic headache after mild head injury: a descriptive study. Cephalalgia. 2014 Mar;34(3):191-200. doi: 10.1177/0333102413505236. Epub 2013 Sep 17. PMID 24045573
- [Background] Rendas-Baum R, Yang M, Varon SF, Bloudek LM, DeGryse RE, Kosinski M. Validation of the Headache Impact Test (HIT-6) in patients with chronic migraine. Health Qual Life Outcomes. 2014 Aug 1;12:117. doi: 10.1186/s12955-014-0117-0. PMID 25080874
- [Background] Yang M, Rendas-Baum R, Varon SF, Kosinski M. Validation of the Headache Impact Test (HIT-6) across episodic and chronic migraine. Cephalalgia. 2011 Feb;31(3):357-67. doi: 10.1177/0333102410379890. Epub 2010 Sep 6. PMID 20819842
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] von Steinbuchel N, Wilson L, Gibbons H, Hawthorne G, Hofer S, Schmidt S, Bullinger M, Maas A, Neugebauer E, Powell J, von Wild K, Zitnay G, Bakx W, Christensen AL, Koskinen S, Formisano R, Saarajuri J, Sasse N, Truelle JL; QOLIBRI Task Force. Quality of Life after Brain Injury (QOLIBRI): scale validity and correlates of quality of life. J Neurotrauma. 2010 Jul;27(7):1157-65. doi: 10.1089/neu.2009.1077. PMID 20210602
- [Background] Lee JJ, Lee MK, Kim JE, Kim HZ, Park SH, Tae JH, Choi SS. Pain relief scale is more highly correlated with numerical rating scale than with visual analogue scale in chronic pain patients. Pain Physician. 2015 Mar-Apr;18(2):E195-200. PMID 25794219
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Provost JS, Petrides M, Monchi O. Dissociating the role of the caudate nucleus and dorsolateral prefrontal cortex in the monitoring of events within human working memory. Eur J Neurosci. 2010 Sep;32(5):873-80. doi: 10.1111/j.1460-9568.2010.07333.x. Epub 2010 Aug 16. PMID 20722715
- [Background] Kashluba S, Casey JE, Paniak C. Evaluating the utility of ICD-10 diagnostic criteria for postconcussion syndrome following mild traumatic brain injury. J Int Neuropsychol Soc. 2006 Jan;12(1):111-8. doi: 10.1017/S1355617706060036. PMID 16433950
- [Background] Olesen, J. Section 5.2.2 Persistent headache attributed to mild traumatic injury to the head. IHS Classification ICHD-3 beta (2016). <https://www.ichd-3.org/5-headache-attributed-to-trauma-or-injury-to-the-head-andor-neck/5-2-persistent-headache-attributed-to-traumatic-injury-to-the-head/5-2-2-persistent-headache-attributed-to-mild-traumatic-injury-to-the-head/>.
- [Derived] Stilling J, Paxman E, Mercier L, Gan LS, Wang M, Amoozegar F, Dukelow SP, Monchi O, Debert C. Treatment of Persistent Post-Traumatic Headache and Post-Concussion Symptoms Using Repetitive Transcranial Magnetic Stimulation: A Pilot, Double-Blind, Randomized Controlled Trial. J Neurotrauma. 2020 Jan 15;37(2):312-323. doi: 10.1089/neu.2019.6692. Epub 2019 Nov 8. PMID 31530227